CLINICAL TRIAL: NCT01422213
Title: Randomised, Double-blind, Parallel-group, Placebo-controlled, Fixed Dose Study on the Efficacy of [Vortioxetine] Lu AA21004 on Cognitive Dysfunction in Adult Patients With Major Depressive Disorder (MDD)
Brief Title: Efficacy Study of Vortioxetine on Cognitive Dysfunction in Adult Patients With Major Depressive Disorder
Acronym: FOCUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14122A; 2011-001572-19 (EudraCT Number)
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-07

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Cognitive dysfunction
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Vortioxetine 10 mg (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)
- Vortioxetine 20 mg (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)

INTERVENTIONS:
Drug: Placebo — capsules; daily; orally
  Arms: Placebo
Drug: Vortioxetine (Lu AA21004) — encapsulated tablets; daily; orally
  Other Names: Brintellix
  Arms: Vortioxetine 10 mg
Drug: Vortioxetine (Lu AA21004) — encapsulated tablets; daily; orally
  Other Names: Brintellix
  Arms: Vortioxetine 20 mg

SUMMARY:
Major Depressive Disorder (MDD) is a severe and common psychiatric disorder. Although MDD primarily involves mood disturbances, patients also usually present alterations in cognitive function (attention, memory, executive functioning and psychomotor speed). Even though antidepressants are suggested in the literature to potentially improve cognitive dysfunction in patients with MDD to some degree, there is a lack of adequate and well-controlled studies to investigate this effect. This study will evaluate the efficacy, safety and tolerability of a new antidepressant Vortioxetine versus placebo on cognitive dysfunction in adult patients with MDD.

ELIGIBILITY:
Inclusion Criteria:

* The patient is an inpatient in a psychiatric hospital or an outpatient at a psychiatric setting at the time of the study entry.
* The patient is diagnosed with recurrent MDD according to DSM-IV-TR™ criteria (classification code 296.3x). The current Major Depressive Episode (MDE) should be confirmed using the Mini International Neuropsychiatric Interview (MINI).
* The patient has received prescribed treatment for a previous episode of depression.
* The patient has a MADRS total score ≥26.
* The reported duration of the current MDE is at least 3 months.

Exclusion Criteria:

* The patient has a score ≥70 on the DSST (number of correct symbols), or ≥42 on the RAVLT (learning) or ≥14 on the RAVLT (memory) at the Baseline Visit.
* The patient has any current Axis I disorder (DSM-IV-TR™ criteria) other than MDD, confirmed using the MINI.
* The patient has a current diagnosis or history of manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features.
* The patient suffers from personality disorders, mental retardation, pervasive development disorder, attention-deficit/hyperactivity disorder, organic mental disorders, or mental disorders due to a general medical condition (DSM-IV-TR™ criteria).
* The patient has physical, cognitive, or language impairment of such severity as to adversely affect the validity of the data derived from the neuropsychological tests.
* The patient is diagnosed with reading disability (dyslexia).
* The patient is at significant risk of suicide or has a score ≥5 on Item 10 (suicidal thoughts) of the MADRS, or has attempted suicide <6 months prior to the Screening Visit.
* The patient has received electroconvulsive therapy <6 months prior to the Screening Visit.
* The current depressive symptoms are considered by the investigator to have been resistant to 2 adequate antidepressant treatments of at least 6 weeks duration each at the recommended dose.
* The patient has a history of moderate or severe head trauma (for example, loss of consciousness for more than 1 hour) or other neurological disorders or systemic medical diseases that are, in the opinion of the investigator, likely to affect central nervous system functioning.
* The patient has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin, that has not been in remission for >5 years prior to the first drug dose.
* The patient has a clinically significant unstable illness, for example:
* cardiovascular disease
* seizure disorder or encephalopathy
* congestive heart failure
* cardiac hypertrophy
* arrhythmia
* bradycardia (pulse <50 bpm)
* respiratory disease
* hepatic impairment or renal insufficiency
* metabolic disorder
* endocrinological disorder
* gastrointestinal disorder
* haematological disorder
* infectious disorder
* any clinically significant immunological condition
* dermatological disorder
* venereal disease
* The patient has, at the Screening Visit, an abnormal ECG that is, in the investigator's opinion, clinically significant.
* The patient is, in the investigator's opinion, unlikely to comply with the protocol or is unsuitable for any reason.
* The patient has previously been exposed to Vortioxetine.

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Derived] Nohr AK, Lindow M, Forsingdal A, Demharter S, Nielsen T, Buller R, Moltke I, Vitezic M, Albrechtsen A. A large-scale genome-wide gene expression analysis in peripheral blood identifies very few differentially expressed genes related to antidepressant treatment and response in patients with major depressive disorder. Neuropsychopharmacology. 2021 Jun;46(7):1324-1332. doi: 10.1038/s41386-021-01002-9. Epub 2021 Apr 8. PMID 33833401
- [Derived] McIntyre RS, Florea I, Tonnoir B, Loft H, Lam RW, Christensen MC. Efficacy of Vortioxetine on Cognitive Functioning in Working Patients With Major Depressive Disorder. J Clin Psychiatry. 2017 Jan;78(1):115-121. doi: 10.4088/JCP.16m10744. PMID 27780334
- [Derived] McIntyre RS, Lophaven S, Olsen CK. A randomized, double-blind, placebo-controlled study of vortioxetine on cognitive function in depressed adults. Int J Neuropsychopharmacol. 2014 Oct;17(10):1557-67. doi: 10.1017/S1461145714000546. Epub 2014 Apr 30. PMID 24787143

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were selected from psychiatric settings, outpatient clinics, and inpatient hospitals; and recruited via ads (if allowed in the country) or referrals (from general practitioners). A Pre-Randomisation Form completed by the site for each patient was reviewed by the CRO Medical Expert to confirm patient eligibility prior to randomisation.
Pre-assignment Details: Patients were randomised equally (1:1:1) at the Baseline Visit to placebo, vortioxetine 10 mg/day, or vortioxetine 20 mg/day for 8 weeks of double-blind treatment (8-week Core Treatment Period).
Groups:
- Vortioxetine 10 mg; Vortioxetine 20 mg: encapsulated tablets; daily; orally
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Started | 196 | 195 | 207
Completed | 163 | 173 | 178
Not Completed | 33 | 22 | 29
Not completed — Adverse Event | 8 | 7 | 11
Not completed — Lack of Efficacy | 10 | 2 | 2
Not completed — Non-compliance with study drug | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 2 | 4
Not completed — Withdrawal of Consent | 7 | 3 | 5
Not completed — Lost to Follow-up | 3 | 3 | 5
Not completed — Administrative or Other Reason(s) | 5 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Age + Gender: all-patients-treated set (APTS) - all patients in the APRS who took at least one dose of IMP.
  Study-specific Measures: full-analysis set (FAS) - all patients in the APTS who had a valid baseline assessment and at least one valid post-baseline assessment of the DSST, RAVLT (learning [acquisition]), and RAVLT (memory [delayed recall]).
Groups:
- Placebo: capsules, daily, orally
- Vortioxetine 10 mg; Vortioxetine 20 mg: encapsulated tablets, daily, orally
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg | Total
Number analyzed (Participants) | 196 | 195 | 207 | 598
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (12.1) | 45.4 (12.2) | 46.1 (11.8) | 45.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 134 | 133 | 396
  Male | 67 | 61 | 74 | 202
DSST: Baseline Total Score [Mean (Standard Deviation); unit: units on a scale] — Digit Symbol Substitution Test (DSST) is a cognitive test designed to assess psychomotor speed of performance requiring visual perception, spatial decision-making, and motor skills. It consists of 133 digits and requires the patient to substitute each digit with a simple symbol in a 90-second period. Each correct symbol is counted, and the total score ranges from 0 (less than normal functioning) to 133 (greater than normal functioning).
  units on a scale | 42.38 (13.76) | 41.96 (12.56) | 41.61 (12.72) | 41.98 (13.00)
RAVLT: Baseline Total Score [Mean (Standard Deviation); unit: correct words] — Rey Auditory Verbal Learning Task (RAVLT) is a cognitive test designed to assess verbal learning and memory, including immediate memory, efficiency of learning, retroactive and proactive interference effects, and encoding versus retrieval. It consists of a number of tasks, including immediate recall and delayed recall. The number of words correctly recalled on each task is recorded. The number of correct words could range from 0 to 45. No categorization of the number of correct words is possible.
  correct words | 22.14 (5.70) | 22.34 (5.76) | 22.64 (5.88) | 22.38 (5.77)
TMT A: Baseline Total Score [Mean (Standard Deviation); unit: seconds] — Trail Making Test (TMT) is a cognitive test designed to assess scanning, visuomotor tracking, executive function, and cognitive flexibility. It consists of two parts, A and B: the patient must draw lines to connect consecutively numbered circles (part A) and then connect consecutively numbered and lettered circles alternating between the two sequences (part B). The time taken to complete the two parts is recorded. Part A assesses cognitive processing speed. The lower the score the faster the processing speed.
  seconds | 48.71 (24.73) | 46.51 (24.12) | 46.23 (26.66) | 47.13 (25.20)
TMT B: Baseline Total Score [Mean (Standard Deviation); unit: seconds] — TMT is a cognitive test designed to assess scanning, visuomotor tracking, executive function, and cognitive flexibility. It consists of two parts, A and B: the patient must draw lines to connect consecutively numbered circles (part A) and then connect consecutively numbered and lettered circles alternating between the two sequences (part B). The time taken to complete the two parts is recorded. Part B examines executive functioning and ability to shift cognitive set. The lower the score the faster the ability to shift cognitive set.
  seconds | 105.05 (52.99) | 101.82 (51.68) | 102.94 (52.43) | 103.27 (52.30)
STROOP Congruent: Baseline Total Score [Mean (Standard Deviation); unit: seconds] — Stroop Colour Naming Test (STROOP) is a cognitive test designed to assess the ability to inhibit a prepotent response to reading words while performing a task that requires attention control. It comprises two sheets with 50 words on each, and each word is the name of a colour. On the Congruent STROOP Sheet, the word and ink colour match; on the Incongruent STROOP Sheet, the word and ink colour do not match. The patient has 4 minutes to name the ink colour of each word. The clinician notes the time taken and counts the number of correct and incorrect responses.
  seconds | 49.97 (24.86) | 49.59 (24.65) | 50.01 (27.58) | 49.86 (25.72)
STROOP Incongruent: Baseline Total Score [Mean (Standard Deviation); unit: seconds] | 85.66 (39.15) | 85.03 (41.09) | 83.62 (41.40) | 84.75 (40.51)
SRT: Baseline Total Score [Mean (Standard Deviation); unit: log10 (ms)] — Simple Reaction Time (SRT) is designed to assess psychomotor speed, and Choice Reaction Time (CRT) is designed to assess visual attention. Two computerised tests, part of the CogState battery were used to measure SRT and CRT in milliseconds:
  * The "detection task" measures SRT: the patient presses a "yes" button, whenever an onscreen playing card is turned over.
  * The "identification task" measures CRT: the patient presses a "yes" button whenever an onscreen playing card is turned over and is red, or a "no" button if the card is not red.
  log10 (ms) | 2.64 (0.20) | 2.64 (0.20) | 2.63 (0.20) | 2.64 (0.20)
CRT: Baseline Total Score [Mean (Standard Deviation); unit: log10 (ms)] — SRT is designed to assess psychomotor speed, and CRT is designed to assess visual attention. Two computerised tests, part of the CogState battery were used to measure SRT and CRT in milliseconds:
  * The "detection task" measures SRT: the patient presses a "yes" button, whenever an onscreen playing card is turned over.
  * The "identification task" measures CRT: the patient presses a "yes" button whenever an onscreen playing card is turned over and is red, or a "no" button if the card is not red.
  log10 (ms) | 2.78 (0.14) | 2.78 (0.14) | 2.78 (0.14) | 2.78 (0.14)
MADRS: Baseline Total Score [Least Squares Mean (Standard Deviation); unit: units on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
  units on a scale | 31.34 (3.75) | 31.62 (3.77) | 31.74 (3.53) | 31.57 (3.68)
CGI-S: Baseline Total Score [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
  units on a scale | 4.55 (0.63) | 4.60 (0.62) | 4.62 (0.58) | 4.59 (0.61)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in DSST (Number of Correct Symbols) and RAVLT (Acquisition and Delayed Recall) Using the Composite Z-score Defined as the Weighted Sum of the Individual Patient Z-scores
Description: DSST assesses psychomotor speed of performance requiring visual perception, spatial decision-making, and motor skills. It consists of 133 digits and requires the patient to substitute each digit with a simple symbol in a 90-s period. Each correct symbol is counted, and the total score ranges from 0 (< normal functioning) to 133 (> normal functioning).
  RAVLT assesses verbal learning and memory, including immediate memory, efficiency of learning, retroactive and proactive interference effects, and encoding versus retrieval. It consists of a number of tasks, including immediate recall and delayed recall. The number of words correctly recalled on each task is recorded.
  The scores are standardized by subtracting the overall mean change from baseline from the individual change from baseline and dividing by the standard deviation estimate of the change from baseline. The 2 tests, DSST and RAVLT are each assigned a weight of 0.5, the 2 subtests of RAVLT are each assigned a weight of 0.25.
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: z score
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 178 | 180 | 187
z score | -0.235 (0.053) | 0.128 (0.052) | 0.095 (0.051)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the composite z-score was analysed using the mixed model for repeated measurements (MMRM) with an unstructured covariance structure. The model included terms for grouped site, baseline composite z-score, baseline composite z-score-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — To adjust for multiplicity, the 10 and 20 mg doses of vortioxetine were tested separately versus placebo in the primary and key secondary efficacy analyses at a Bonferroni-corrected significance level of 0.05/2 = 0.025; Mean Difference (Final Values) = 0.363, 95% CI 2-sided [0.22 to 0.50], Standard Error of Mean 0.072
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Based on the FAS, the composite z-score was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site, baseline composite z-score, baseline composite z-score-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.330, 95% CI 2-sided [0.19 to 0.47], Standard Error of Mean 0.071

2. Secondary Outcome: Change From Baseline to Week 8 in DSST (Number of Correct Symbols)
Description: Digit Symbol Substitution Test (DSST) is a cognitive test designed to assess psychomotor speed of performance requiring visual perception, spatial decision-making, and motor skills. It consists of 133 digits and requires the patient to substitute each digit with a simple symbol in a 90-second period. Each correct symbol is counted, and the total score ranges from 0 (less than normal functioning) to 133 (greater than normal functioning)." as a description of DSST.
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: number of correct symbols
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 179 | 180 | 187
number of correct symbols | 4.83 (0.63) | 9.03 (0.63) | 9.09 (0.61)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the DSST (number of correct symbols) was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site, baseline value, baseline value-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.20, 95% CI 2-sided [2.50 to 5.90], Standard Error of Mean 0.87
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.26, 95% CI 2-sided [2.57 to 5.94], Standard Error of Mean 0.86

3. Secondary Outcome: Change From Baseline to Week 8 in RAVLT (Acquisition)
Description: Rey Auditory Verbal Learning Task (RAVLT) is a cognitive test designed to assess verbal learning and memory, including immediate memory, efficiency of learning, retroactive and proactive interference effects, and encoding versus retrieval. It consists of a number of tasks, including immediate recall and delayed recall. The number of words correctly recalled on each task is recorded.
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: number of words correctly recalled
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 179 | 180 | 187
number of words correctly recalled | 3.06 (0.34) | 4.08 (0.34) | 3.65 (0.33)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the RAVLT (acquisition) was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site, baseline value, baseline value-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p = 0.0287, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.02, 95% CI 2-sided [0.11 to 1.93], Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1988, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [-0.31 to 1.50], Standard Error of Mean 0.46

4. Secondary Outcome: Change From Baseline to Week 8 in RAVLT (Delayed Recall)
Description: as for outcome 3
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: number of words correctly recalled
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 178 | 180 | 187
number of words correctly recalled | 0.91 (0.18) | 1.63 (0.18) | 1.56 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the RAVLT (delayed recall) was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site, baseline value, baseline value-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p = 0.0033, Mixed Models Analysis — Since the p-value for RAVLT acquisition for 10 mg was >0.025, the p-value for this test is nominal; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [0.24 to 1.19], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0073, Mixed Models Analysis — Since the p-value for RAVLT acquisition for 20 mg was >0.025, the p-value for this test is nominal; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [0.17 to 1.12], Standard Error of Mean 0.24

5. Secondary Outcome: Change From Baseline to Week 8 in the TMT A (Speed of Processing)
Description: Trail Making Test (TMT) is a cognitive test designed to assess scanning, visuomotor tracking, executive function, and cognitive flexibility. It consists of two parts, A and B: the patient must draw lines to connect consecutively numbered circles (part A) and then connect consecutively numbered and lettered circles alternating between the two sequences (part B). The time taken to complete the two parts is recorded. Part A assesses cognitive processing speed. The lower the score the faster the processing speed.
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 179 | 180 | 187
seconds | -7.07 (1.00) | -10.84 (1.00) | -10.87 (0.97)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the TMT A (Speed of Processing) was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site, baseline value, baseline value-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p = 0.0061, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -3.76, 95% CI 2-sided [-6.45 to -1.08], Standard Error of Mean 1.37
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0052, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -3.80, 95% CI 2-sided [-6.46 to -1.14], Standard Error of Mean 1.35

6. Secondary Outcome: Change From Baseline to Week 8 in the TMT B (Executive Function)
Description: TMT is a cognitive test designed to assess scanning, visuomotor tracking, executive function, and cognitive flexibility. It consists of two parts, A and B: the patient must draw lines to connect consecutively numbered circles (part A) and then connect consecutively numbered and lettered circles alternating between the two sequences (part B). The time taken to complete the two parts is recorded. Part B examines executive functioning and ability to shift cognitive set. The lower the score the faster the ability to shift cognitive set.
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 179 | 180 | 186
seconds | -13.84 (2.00) | -21.41 (2.00) | -22.85 (1.95)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the TMT B (Executive Function) was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site, baseline value, baseline value-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p = 0.0058, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -7.57, 95% CI 2-sided [-12.93 to -2.20], Standard Error of Mean 2.73
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -9.01, 95% CI 2-sided [-14.32 to -3.70], Standard Error of Mean 2.70

7. Secondary Outcome: Change From Baseline to Week 8 in Congruent STROOP Time to Complete (Executive Function)
Description: Stroop Colour Naming Test (STROOP) is a cognitive test designed to assess the ability to inhibit a prepotent response to reading words while performing a task that requires attention control. It comprises two sheets with 50 words on each, and each word is the name of a colour. On the first sheet, the Congruent STROOP Sheet, the word and ink colour match; on the Incongruent STROOP Sheet, the word and ink colour do not match. For each sheet, the patient has 4 minutes to name the ink colour of each word. When the patient finishes the sheet, or once 4 minutes is up, the clinician notes the time taken and counts the number of correct and incorrect responses. The scale ranges from 0-100, the higher score the greater the cognitive flexibility.
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 179 | 180 | 186
seconds | -5.97 (0.93) | -9.97 (0.93) | -10.43 (0.90)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the Congruent STROOP Time to Complete (Executive Function) was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site, baseline value, baseline value-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -4.00, 95% CI 2-sided [-6.50 to -1.49], Standard Error of Mean 1.28
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -4.45, 95% CI 2-sided [-6.93 to -1.97], Standard Error of Mean 1.26

8. Secondary Outcome: Change From Baseline to Week 8 in Incongruent STROOP Time to Complete (Executive Function)
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 176 | 178 | 184
seconds | -10.94 (1.48) | -17.69 (1.48) | -17.45 (1.44)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the Incongruent STROOP Time to Complete (Executive Function) was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site, baseline value, baseline value-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -6.75, 95% CI 2-sided [-10.76 to -2.74], Standard Error of Mean 2.04
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -6.52, 95% CI 2-sided [-10.49 to -2.54], Standard Error of Mean 2.02

9. Secondary Outcome: Change From Baseline to Week 8 in the SRT (Speed of Processing)
Description: Simple Reaction Time (SRT) is designed to assess psychomotor speed, and Choice Reaction Time (CRT) is designed to assess visual attention. Two computerised tests, part of the CogState battery were used to measure SRT and CRT in milliseconds:
  * The "detection task" measures SRT: the patient presses a "yes" button, whenever an onscreen playing card is turned over.
  * The "identification task" measures CRT: the patient presses a "yes" button whenever an onscreen playing card is turned over and is red, or a "no" button if the card is not red.
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: log10 (ms)
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 169 | 176 | 176
log10 (ms) | -0.007 (0.009) | -0.053 (0.009) | -0.037 (0.009)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the SRT (Speed of Processing) was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site, baseline value, baseline value-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -0.046, 95% CI 2-sided [-0.07 to -0.02], Standard Error of Mean 0.012
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0157, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -0.029, 95% CI 2-sided [-0.05 to -0.01], Standard Error of Mean 0.012

10. Secondary Outcome: Change From Baseline to Week 8 in the CRT (Attention)
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: log10 (ms)
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 169 | 176 | 180
log10 (ms) | -0.015 (0.007) | -0.046 (0.007) | -0.023 (0.006)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the CRT (Attention) was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site, baseline value, baseline value-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -0.032, 95% CI 2-sided [-0.05 to -0.01], Standard Error of Mean 0.009
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.3549, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.03 to 0.01], Standard Error of Mean 0.009

11. Secondary Outcome: Change From Baseline to Week 8 in MADRS Total Score
Description: The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 165 | 174 | 181
units on a scale | -10.85 (0.64) | -15.56 (0.63) | -17.55 (0.62)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the MADRS Total Score was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site, baseline value, baseline value-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -4.70, 95% CI 2-sided [-6.45 to -2.96], Standard Error of Mean 0.89
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -6.70, 95% CI 2-sided [-8.43 to -4.98], Standard Error of Mean 0.88

12. Secondary Outcome: Change From Baseline to Week 8 in CGI-S Score
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 165 | 174 | 181
units on a scale | -1.15 (0.08) | -1.80 (0.08) | -2.00 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the CGI-S Score was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site, baseline value, baseline value-by-visit interaction, and treatment-by-visit interaction; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-0.88 to -0.42], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-1.08 to -0.62], Standard Error of Mean 0.12

13. Secondary Outcome: Clinical Status Using CGI-I Score at Week 8
Description: The Clinical Global Impression - Global Improvement (CGI-I) is a 7-point scale rated from 1 (very much improved) to 7 (very much worse). The investigator rated the patient's overall improvement relative to baseline, whether or not, in the opinion of the investigator, this was entirely due to the drug treatment.
Time Frame: Week 8
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 165 | 174 | 181
units on a scale | 2.85 (0.08) | 2.24 (0.08) | 1.99 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Based on the FAS, the CGI-I Score was analysed using the MMRM with an unstructured covariance structure. The model included terms for grouped site and treatment-by-visit interaction; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.81 to -0.40], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — No adjustment for multiplicity was made; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-1.06 to -0.65], Standard Error of Mean 0.11

14. Secondary Outcome: Proportion of Responders at Week 8 (Response Defined as a >=50% Decrease in the MADRS Total Score From Baseline
Time Frame: Baseline and Week 8
Population: FAS, last observation carried forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 194 | 193 | 204
percentage of participants | 29.4 | 47.7 | 58.8
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.0002, Regression, Logistic — Wald's Test. No adjustment for multiplicity was made; Odds Ratio (OR) = 2.19, 95% CI 2-sided [1.44 to 3.33]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Wald's Test. No adjustment for multiplicity was made; Odds Ratio (OR) = 3.43, 95% CI 2-sided [2.26 to 5.21]

15. Secondary Outcome: Proportion of Remitters at Week 8 (Remission is Defined as a MADRS Total Score <=10)
Time Frame: Week 8
Population: FAS, LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 194 | 193 | 204
percentage of participants | 17.0 | 29.5 | 38.2
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.0030, Regression, Logistic — Wald's Test. No adjustment for multiplicity was made; Odds Ratio (OR) = 2.09, 95% CI 2-sided [1.29 to 3.41]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Wald's Test. No adjustment for multiplicity was made; Odds Ratio (OR) = 3.13, 95% CI 2-sided [1.95 to 5.03]

16. Secondary Outcome: Change From Baseline to Week 1 Using the MADRS Total Score and the Composite Z-score
Description: Effect on cognitive dysfunction after correcting for the effect on depressive symptoms.
  The estimation of the effect on cognitive dysfunction after correcting for the effect on depressive symptoms was based on the composite z-score and the MADRS total score. The effect was estimated in an ANCOVA model using the composite z-score at week 1 as dependent variable and the change from baseline to week 1 in the MADRS total score, the baseline MADRS total score, the baseline composite z-score, the treatment group and site as independent variables.
  In the week 1 analysis the vortioxetine 10 and 20 mg groups were pooled because patients randomized to vortioxetine 20 mg received vortioxetine 10 mg in the first week of the study.
Time Frame: Baseline and Week 1
Population: FAS, LOCF
Measure: Least Squares Mean (Standard Error); unit: z score
Arm/Group | Placebo | Vortioxetine 10 mg
Number analyzed (Participants) | 193 | 389
z score | -0.079 (0.050) | 0.042 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.0393, ANCOVA — No adjustment for multiplicity was made; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.01 to 0.24], Standard Error of Mean 0.059

17. Secondary Outcome: Change From Baseline to Week 8 Using the MADRS Total Score and the Composite Z-score
Description: Effect on cognitive dysfunction after correcting for the effect on depressive symptoms.
  The estimation of the effect on cognitive dysfunction after correcting for the effect on depressive symptoms was based on the composite z-score and the MADRS total score. The effect was estimated in an ANCOVA model using the composite z-score at week 1 as dependent variable and the change from baseline to week 1 in the MADRS total score, the baseline MADRS total score, the baseline composite z-score, the treatment group and site as independent variables.
Time Frame: Baseline and Week 8
Population: FAS, LOCF
Measure: Least Squares Mean (Standard Error); unit: z score
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 194 | 193 | 204
z score | -0.189 (0.050) | 0.041 (0.049) | -0.036 (0.048)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.0007, ANCOVA — No adjustment for multiplicity was made; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [0.10 to 0.36], Standard Error of Mean 0.068
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority or Other; p = 0.0246, ANCOVA — No adjustment for multiplicity was made; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.02 to 0.29], Standard Error of Mean 0.068

18. Secondary Outcome: Risk of Suicidality Using C-SSRS Scores
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) was developed by researchers at Columbia University as a tool to systematically assess suicidal ideation and behaviour in patients during participation in a clinical study. The C-SSRS is composed of questions that address suicidal behaviour and questions that address suicidal ideation, with subquestions that assess severity. The tool was administered via an interview with the patient.
  For 2 patients in each treament group (6 in total) the CSSRS assessments are missing during study.
Time Frame: Up to 8 weeks
Population: APTS
Measure: Number; unit: participants
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 196 | 195 | 207
participants
  No suicidal ideation or behaviour | 173 | 175 | 178
  Any non-suicidal self-injurious behavior | 0 | 0 | 0
  Any suicidal ideation or behaviour | 21 | 18 | 27

ADVERSE EVENTS:
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Serious Adverse Events (participants affected / at risk) | 2/196 | 0/195 | 2/207
Other Adverse Events (participants affected / at risk) | 31/196 | 48/195 | 66/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=196) | Vortioxetine 10 mg (N=195) | Vortioxetine 20 mg (N=207)
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=196) | Vortioxetine 10 mg (N=195) | Vortioxetine 20 mg (N=207)
Nausea (Gastrointestinal disorders) | 8 | 32 | 43
Nasopharyngitis (Infections and infestations) | 10 | 7 | 9
Headache (Nervous system disorders) | 14 | 16 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study will be published. Authors of the primary publication based on this study must fulfil the criteria defined by the International Committee of Medical Journal Editors (ICMJE). The primary publication must be published before any secondary publications are submitted for publication.